CLINICAL TRIAL: NCT05810415
Title: Use of Renin Versus Lactic Acid as Tissue Perfusion Biomarkers for Mortality Prediction in Hypotensive Critically Ill Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, mohamed A Aboelsuod, MD, assistant professor of anesthesia intensive care and pain management, Al-Azhar University
Other Study IDs: 221190
Record Dates: First submitted 2023-01-21; First posted 2023-04-12 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Sepsis; Obstructive Shock; Critical Illness; Hypotensive; Critically Ill
MeSH Terms: conditions — Sepsis; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Renin group and lactate group: Renin group and lactate group
  Interventions: Diagnostic Test: Renin levels and lactic acid levels

INTERVENTIONS:
Diagnostic Test: Renin levels and lactic acid levels — Sampling of blood for measuring renin and lactate

SUMMARY:
Measurement of Whole Blood Lactate Concentrations Whole blood lactate concentrations will be measured at the time of study enrollment and at 24, 48, and 72 hours. Measurement of Plasma Renin Concentrations Serum renin concentration will be measured on blood samples drawn from arterial catheters on supine position right after inclusion. Discarded whole blood samples (waste blood samples) in EDTA tubes are prospectively collected from each patient at the time of study enrollment and at 24, 48, and 72 hours.

DETAILED DESCRIPTION:
Elevated renin-levels in critically ill patients are associated with worse outcomes and outperform lactate as a prognostic indicator of survival. Using biomarkers to understand patient trajectory in the ICU has high utility.

Both whole blood lactate concentration and lactate clearance yield meaningful information, but lactate can be an insensitive prognostic marker. Renin has recently emerged as a prognostic marker for ICU mortality.

AIM OF THE WORK Evaluation of serum renin level to determine if it performs well as a marker of tissue-perfusion and prediction of mortality of critically ill patients in intensive care unit in comparison with serum lactate.

a prospective observational study will be conducted.. Patients can be enrolled at any point during their admission. The patients are followed once enrolled and the data are recorded till death or end of ICU stay by dedicated investigator. Primary and secondary outcomes will be analyzed after completing of the study.

Plasma renin concentrations and Whole blood lactate concentrations are measured at enrollment and at 24, 48, and 72 hours.

Measurements

1. Patient characteristics: including age, sex, chronic health conditions, weight.
2. Reasons of ICU admission.
3. length of stay in days (ICU and hospital).
4. Mortality (ICU and in-hospital).
5. Physiologic data: including heart rate, mean arterial blood pressure (MAP), temperature, respiratory rate, PaO2, FIO2, hematocrit, WBC count, serum creatinine, urine output, blood urea nitrogen, sodium, albumin, bilirubin, glucose, arterial carbon dioxide tension, pH, and the total Glasgow Coma Scale score.
6. The need for mechanical ventilation and renal replacement therapy.
7. Patient outcome either survivor or not survivor. Measurement of Whole Blood Lactate Concentrations Whole blood lactate concentrations will be measured at the time of study enrollment and at 24, 48, and 72 hours.

Measurement of Plasma Renin Concentrations Serum renin concentration will be measured on blood samples drawn from arterial catheters on supine position right after inclusion.

Discarded whole blood samples (waste blood samples) in EDTA tubes are prospectively collected from each patient at the time of study enrollment and at 24, 48, and 72 hours.

Samples will be centrifuged to yield 2mL of EDTA plasma and then stored at -20°C. After all samples for the study are collected, frozen samples are thawed for batch analysis.

Plasma active renin levels are measured using the active renin enzyme-linked immunosorbent assay kit.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 21-60 years old
2. Those receiving vasopressors for greater than or equal to 6 hours to maintain a mean arterial pressure (MAP) ≥65 mm Hg.
3. Anticipated stay >24 hours.

Exclusion Criteria:

1. Patients or families refusing to participate in the study.
2. Patients on renal replacement therapy.
3. Patients receiving betablockers

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study will be conducted at Al-Azhar university hospitals at intensive care unit (ICU). Patients can be enrolled at any point during their admission. The patients are followed once enrolled and the data are recorded till death or end of ICU stay by dedicated investigator
Sampling Method: Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2022-06-21 (Actual); Primary Completion 2024-01-25 (Estimated); Study Completion 2024-01-25 (Estimated)

PRIMARY OUTCOMES:
Evaluation of serum renin level as a marker of tissue perfusion and prediction of mortality of critically ill patients in intensive care unit in comparison with serum lactate. | from baseline to 72 hours after enrollment to intensive care unit (ICU)
  Number of HYPOTENSIVE CRITICALLY ILL PATIENTS through measurements of the Plasma renin concentrations and Whole blood lactate concentrations at enrollment to intensive care unit (ICU) and at 24, 48, and 72 hours after enrollment

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Azhar University, Madīnat an Naşr, Cairo Governorate
  - Azhar unversity, Cairo

IPD SHARING:
Plan to Share IPD: Undecided